CLINICAL TRIAL: NCT05361018
Title: SensiEx - Sensorimotor Training Using Whole Body Vibration Exercise to Reduce Chemotherapy-induced Peripheral Neuropathy After Treatment for Breast Cancer a Randomized Controlled Pilot Trial
Brief Title: Sensorimotor Training Using Whole Body Vibration Exercise to Reduce Chemotherapy-induced Peripheral Neuropathy
Acronym: Sensi-Ex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Yvonne Wengstrom, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Yvonne Wengstrom
Record Dates: First submitted 2022-04-11; First posted 2022-05-04 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Breast Neoplasm, Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: two-armed, randomized controlled design. Patients will then be assigned randomly either to the WBV group or the CAR group. Patients allocated to the WBV group receive a defined WBV exercise program twice a week in addition to their usual treatment. Patients in conventional aerobic and resistance exercise (CAR) group will receive a defined exercise program twice a week in addition to their usual treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Body Vibration exercise - WBV (Experimental): The vibration exercises take place on a tri-planar vibration platform (Power Plate) according to the initially determined setting for each individual (highest, though feasible neuromuscular response). . Each session lasts for about 15-30 min in total, leaving sufficient time for regeneration. Training consists of at least four vibration exercises, chosen from a standardized pool of exercises with increasing difficulty in order to allow for individual, optimal progression. All sessions and adherence are documented by the exercise supervisor. Adverse events are documented, and patients asked to give feedback regarding the feasibility and subjective impression of each individual setting. All training sessions will be supervised. The participants rating of perceived exertion (RPE) will be assessed immediately after each set of exercise.
  Interventions: Other: Whole Body Vibration exercise - WBV
- Conventional Aerobic and Resistance exercise - CAR (Active Comparator): exercise sessions commence with 20 min of moderate intensity continuous aerobic exercise at a rating of perceived exertion (RPE) of 13-15 on the Borg scale. Participants complete both resistance exercises and high intensity intermittent aerobic exercises during each session. The resistance training regimen consists of 8 exercises (leg press, biceps curls, triceps extensions, bench press, shoulder press, standing row, sit ups/Russian weighted abdominal twist, and prone lying back extensions. Participants complete 2 sets of 8-12 repetitions at an initial intensity of 70 % of their estimated 1 repetition maximum (1-RM) strength and increase to 80 % of estimated 1-RM when more than 12 repetitions can be correctly performed by the participant
  Interventions: Other: Whole Body Vibration exercise - WBV

INTERVENTIONS:
Other: Whole Body Vibration exercise - WBV — participants will be randomised to two different training interventions
  Other Names: Conventional Aeorbic and Resistance exercise - CAR

SUMMARY:
CIPN is induced by neurotoxic chemotherapeutic agents and manifests with sensory and/or motor deficits. It is associated with significant disability and poor recovery. Common symptoms include pain, altered sensation, reduced or absent reflexes, muscle weakness, reduced balance control and insecure gait. The purpose of the study is to compare effects of sensory vibrations training to conventional aerobic and strenght exercise on neurophatic symptoms related to chemotherapy treatment.

DETAILED DESCRIPTION:
Aim: To (a) compare the effects of WBV exercise compared to regular cardiovascular and resistance exercise (CAR) on the primary outcome of (a) CIPN symptoms and secondary outcomes of (b) balance, physical function, and quality of life.

Based on previous pilot study findings, we hypothesize that WBV exercise compared to CAR will reduce relevant symptoms to a larger degree, such as the loss of peripheral deep sensitivity, pain, weakened or absent reflexes and loss of balance control (aim a) and that patients will experience an improvement in physical function and quality of life (aim b).

The study employs a prospective, multicenter, two-armed, randomized controlled design. Study participants will be informed about the study procedure and sign a written informed consent. Patients will then be assigned randomly either to the WBV group or the CAR group. Patients allocated to the WBV group receive a defined WBV exercise program twice a week in addition to their usual treatment. Patients in conventional aerobic and resistance exercise (CAR) group will receive a defined exercise program twice a week in addition to their usual treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with breast cancer, aged 18-80 years,
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2,
* completed chemotherapy in the past 3 months. Experiencing symptoms of CIPN

Exclusion Criteria:

* pre-existing neuropathy of other cause (eg, diabetes),
* given contraindications for WBV including instable bone metastases and severe cardiovascular disease.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Chemotherapy-induced peripheral neuropathy subjective symptoms, less symptoms | Change from Baseline to 12 weeks
  Chemotherapy-induced peripheral neuropathy assessed by The Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) symptom experience scale
Chemotherapy-induced peripheral neuropathy sensory loss assessment, increased sensation | Change from Baseline to 12 weeks
  Monofilament testing will be performed to further quantify sensory loss at all three time points by a specially trained researcher with Von Frey Monofilament Kit using established procedures by Dyck and colleagues

SECONDARY OUTCOMES:
Balance control, improved balance | Change from Baseline to12 weeks
  Unipedal Stance Time test
Performance status, improved balance and function | Change from Baseline to 12 weeks
  Timed Up and Go (TUG)
Additional balance assessment | Change from Baseline to 12 weeks
  Modified Clinical Test for Sensory Interaction in Balance (mCTSIB)
Pain related to CIPN, less pain than baseline | Change from Baseline to 12 weeks
  The painDETECT questionnaire
Quality of Life assessment, improved quality of life | Change from Baseline to 12 weeks
  The EORTC-QLQ-C30 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Wengström, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No